CLINICAL TRIAL: NCT04595279
Title: Cigarette Smoking Decision Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IRB00264306; R01DA049814 (NIH)
Record Dates: First submitted 2020-10-14; First posted 2020-10-20 (Actual); Results first posted 2025-06-15 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-05

CONDITIONS: Tobacco Smoking
MeSH Terms: conditions — Tobacco Smoking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Smoking sessions (Experimental): This is the single arm that will go through cigarette smoking sessions
  Interventions: Behavioral: Smoking sessions

INTERVENTIONS:
Behavioral: Smoking sessions — Participants undergo topography and behavioral economic sessions where they can make choices to earn cigarette puffs by pulling plungers on experimental equipment

SUMMARY:
The Family Smoking Prevention and Tobacco Control Act granted the FDA the authority to regulate and restrict tobacco advertising tactics that inaccurately convey reduced product risk, yet there is a dearth of up-to-date regulatory science to inform such regulations. Although the FDA has restricted use of descriptors such as "natural" and "additive-free," research shows that the tobacco industry quickly pivoted to increase use of alternative, unregulated tactics. Greenwashing is one increasingly common tobacco marketing strategy in which products are portrayed as eco-friendly and/or natural. The investigators' preliminary research indicates that greenwashing tactics may inaccurately convey modified product risk to consumers. The overarching objective of this project is to test the effect of greenwashing methods used by cigarette companies to market products on actual smoking behavior in a controlled laboratory study. The investigators' proposed research focuses on young adults (age 18-29), because this is a key age for smoking initiation and escalation, and research has found that young adults may be more susceptible than older adults to greenwashing in cigarette ads. This study will test the effect of greenwashing on behavioral economic demand and smoking topography in a laboratory-controlled cigarette self-administration study. These data will clearly connect tobacco advertising features to product risk perceptions and actual smoking behavior. This work will provide FDA with an integrated set of evidence that identifies misleading greenwashing tactics that inaccurately convey modified product risk which can be used to inform regulatory action regarding restrictions of this type of advertising.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 29 years of age
* Smoke at least five cigarettes per day
* Have an expired carbon monoxide level of more than 8 ppm or a urinary cotinine level of more than 100 ng per milliliter

Exclusion Criteria:

* The intention to quit smoking in the next 30 days
* Report "roll your own" cigarettes as an exclusive form of smoking
* A serious medical or psychiatric disorder or unstable condition
* Any positive toxicological screening for illicit drugs other than cannabis will be excluded
* Women who are pregnant, plan to become pregnant or are breast-feeding

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2021-08-18 (Actual); Primary Completion 2024-03-22 (Actual); Study Completion 2024-03-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew W Johnson, Ph.D., Principal Investigator — Professor
Locations (1):
- Behavioral Pharmacology Research Unit, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Greenwashing and Control Advertising: This is the single arm that will go through 9 cigarette smoking sessions. Participants complete 9 experimental sessions in which they see concurrently presented greenwashing and control advertisements for cigarettes. Data are from those 9 sessions.
  Smoking sessions: Participants undergo topography and behavioral economic sessions where they can make choices to earn cigarette puffs by pulling plungers on experimental equipment. There is a within-session randomization to earn greenwashing versus control advertised cigarettes. Both conditions were present in each session with variations in cost.
Period: Overall Study
Arm/Group | Greenwashing and Control Advertising
Started | 37
Completed | 31
Not Completed | 6

BASELINE CHARACTERISTICS:
Arm/Group | Smoking Sessions
Number analyzed (Participants) | 37
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.5 (4.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 14
  White | 13
  More than one race | 5
  Unknown or Not Reported | 2

OUTCOME MEASURES:

1. Primary Outcome: Demand Intensity as Assessed by a Behavioral Economic Demand Curve
Description: Number of cigarette puff bouts smoked at no cost as measured by a demand curve
Time Frame: Through study completion, an average of 2 weeks
Population: Participants that completed the study
Measure: Mean (Standard Deviation); unit: puff bouts
Groups:
- Greenwashing and Control Advertising: Participants completed 9 experimental sessions in which they saw concurrently presented greenwashing and control advertisements for cigarettes. Data are from those 9 sessions.
Arm/Group | Greenwashing and Control Advertising
Number analyzed (Participants) | 31
puff bouts
  Greenwashing Advertisment | 4.709677419 (3.588811766)
  Control Advertisement | 2.580645161 (3.442617159)

2. Primary Outcome: Demand Elasticity as Assessed by a Behavioral Economic Demand Curve
Description: Sensitivity of cigarette consumption to changes in cost for cigarettes
Time Frame: Through study completion, an average of 2 weeks
Population: Data could not be summarized for elasticity measures due to lack of non-zero responding at higher prices on the demand curve.
Arm/Group | Greenwashing and Control Advertising
Number analyzed (Participants) | 0

3. Primary Outcome: Cross-price Elasticity Coefficients as Assessed by a Behavioral Economic Demand Curve
Description: Sensitivity of cigarette consumption to changes in cost for alternative products as a linear slope.
Time Frame: Through study completion, an average of 2 weeks
Population: Participants that completed the study
Measure: Mean (Standard Deviation); unit: slope
Arm/Group | Greenwashing and Control Advertising
Number analyzed (Participants) | 31
slope
  Greenwashing Advertising | 0.03 (0.09)
  Control Advertising | 0.05 (0.12)

4. Primary Outcome: Change in Total Puff Volume as Measured by a Smoking Topography Machine
Description: Total cigarette puff volume in milliliters (mls)
Time Frame: Days 2 and 3
Population: Participants that completed the study
Measure: Mean (Standard Error); unit: mLs
Arm/Group | Greenwashing and Control Advertising
Number analyzed (Participants) | 31
mLs
  Greenwashing Advertising | 1649 (1490)
  Control Advertising | 1321 (883.7)

ADVERSE EVENTS:
Time Frame: Up to 2 months
Arm/Group | Smoking Sessions
All-Cause Mortality (participants affected / at risk) | 0/37
Serious Adverse Events (participants affected / at risk) | 0/37
Other Adverse Events (participants affected / at risk) | 0/37

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-02-18): https://cdn.clinicaltrials.gov/large-docs/79/NCT04595279/Prot_SAP_000.pdf